CLINICAL TRIAL: NCT06138522
Title: Qualitative Study on the Perception of Changes in the Psychotherapy of Traumatized Young People
Acronym: TRAUMADOPSY
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231046; 2023-A01689-36 (Other: French Ministry of Health)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Post-traumatic stress disorder; Psychotherapy; Qualitative study
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents: Participants in consultations specialising in the treatment of psychotrauma at the Maison de Solenn
  Interventions: Behavioral: Semi-structured interviews; Behavioral: Child Post-Traumatic Stress Response Index (CPTS-RI) scale; Behavioral: - Therapeutic Alliance Questionnaire (HAQ-CP)
- Parents: Participants in consultations specialising in the treatment of psychotrauma at the Maison de Solenn
  Interventions: Behavioral: Semi-structured interviews; Behavioral: - Therapeutic Alliance Questionnaire (HAQ-CP)
- Professionals: Participants in consultations specialising in the treatment of psychotrauma at the Maison de Solenn
  Interventions: Behavioral: - Therapeutic Alliance Questionnaire (HAQ-CP)

INTERVENTIONS:
Behavioral: Semi-structured interviews — Semi-structured interviews
  Groups: Adolescents; Parents
Behavioral: Child Post-Traumatic Stress Response Index (CPTS-RI) scale — Child Post-Traumatic Stress Response Index (CPTS-RI) scale
  Groups: Adolescents
Behavioral: - Therapeutic Alliance Questionnaire (HAQ-CP) — - Therapeutic Alliance Questionnaire (HAQ-CP)

SUMMARY:
The clinic of psychological trauma in adolescents still requires further development, whereas it is well documented in adults. This clinic is complex, because it must take into account the nature and type of trauma (recent or not, intentional or not, situations of abuse or sexual violence, etc.), the impact on development, the contexts (social, cultural and family) in which the trauma occurs, and the various vulnerability factors associated with it. This complexity has implications for psychotherapeutic management, which needs to be tailored to the specific clinical profiles of adolescents.

Several studies have evaluated psychotherapy for traumatized adolescents, showing a positive short-term effect on the reduction of post-traumatic stress symptoms, whatever the type of psychotherapy. Few studies, however, have analyzed the therapeutic process and the common factors of change, linked mainly to the therapeutic alliance, the patient's experience and the therapist's role: key factors of change according to the international literature. In this context, the patient's experience of his or her psychotherapeutic follow-up is a source of information that has long been neglected, even though it seems essential for better investigating and understanding the complexity of the processes at play in trauma psychotherapy.

DETAILED DESCRIPTION:
The clinic of psychological trauma in adolescents still requires further development, whereas it is well documented in adults. This clinic is complex, because it must take into account the nature and type of trauma (recent or not, intentional or not, situations of abuse or sexual violence, etc.), the impact on development, the contexts (social, cultural and family) in which the trauma occurs, and the various vulnerability factors associated with it. This complexity has implications for psychotherapeutic management, which needs to be tailored to the specific clinical profiles of adolescents.

Several studies have evaluated psychotherapy for traumatized adolescents, showing a positive short-term effect on the reduction of post-traumatic stress symptoms, whatever the type of psychotherapy. Few studies, however, have analyzed the therapeutic process and the common factors of change, linked mainly to the therapeutic alliance, the patient's experience and the therapist's role: key factors of change according to the international literature. In this context, the patient's experience of his or her psychotherapeutic follow-up is a source of information that has long been neglected, even though it seems essential for better investigating and understanding the complexity of the processes at play in trauma psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

Teenagers :

* Teenagers from 12 to 18 years old
* Post-traumatic stress disorder (DSM Criteria 5 Post-Traumatic Stress Disorder)
* Consultant at the Maison de Solenn (Maison des Adolescents)
* Affiliated to a social security scheme

Parents : parents of adolescents followed at the MDA and agreeing to participate in the study

Professionals: providing psychotherapeutic follow-up for adolescents at the MDa

Exclusion Criteria:

* Refusal of the adolescent and/or his/her family (if applicable) to participate in the study,
* Adults (all groups combined): under guardianship or curatorship, under judicial protection

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents suffering from psychotrauma and psychotherapy follow-up in the Consultation Service, Maison de Solenn, Maison des adolescents de l'hôpital Cochin (AP-HP).
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interviews | At the end of the psychotherapy (up to month 12)
  Adolescent Psychotherapy Experience = Evolution in semi-structured interviews at the beginning (T1) and end (T2) of psychotherapy (adolescents)

SECONDARY OUTCOMES:
Child Post-Traumatic Stress Response Index (CPTS-RI) scale | At the end of the psychotherapy (up to month 12)
  Evolution of psychotraumatic symptoms in adolescents (CPTS-IR) between the beginning (T1) and the end of psychotherapy (T2) (adolescents).
  The Child Posttraumatic Stress Reaction Index (CPTS-RI) measures the presence of post-traumatic stress disorder:
  Severity is generally assessed according to the following criteria:
  0 - 11: mild, 11 - 24: mild, 25 - 39: moderate, 40 - 59: severe, 60 - 80: very severe.
Therapeutic Alliance Questionnaire (HAQ-CP) | At the end of the psychotherapy (up to month 12)
  Perception of change, the therapeutic alliance perceived by adolescents, parents and therapists at the end of psychotherapy (adolescents + parents + professionals).
  The Helping Alliance Questionnaires for Child and Parents (HAQ-CP) assesses the quality of the therapeutic alliance.
  Answers to the questionnaires produce 2 scores:
  An alliance score ranging from 0 (weak alliance) to 100 (strong alliance) A well-being score ranging from 0 (feeling unwell) to 10 (feeling well).
Semi-structured interviews | At the end of the psychotherapy (up to month 12)
  Experience at the end (T2) of psychotherapy (parents)

CONTACTS AND LOCATIONS:
Overall Officials: Sevan Minassian, MD, Principal Investigator — University Hospital Cochin, Maison des Adolescents - Youth Department, F-75014 Paris, France
Locations (1):
- University Hospital Cochin, Maison des Adolescents - Youth Department, F-75014 Paris, France, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No